CLINICAL TRIAL: NCT00514345
Title: CYP3A5 Genotype as a Potential Risk Factor for the Development of Ifosamide Nephrotoxicity in Children
Brief Title: CYP3A5 Gene as a Risk Factor for Kidney Damage in Young Patients With Cancer Treated With Ifosfamide
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CCLG-PK-2007-02; CDR0000560128 (Registry Identifier: PDQ (Physician Data Query)); EU-20743
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Chemotherapeutic Agent Toxicity; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: chemotherapeutic agent toxicity; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; nonmetastatic childhood soft tissue sarcoma; unspecified childhood solid tumor, protocol specific; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymorphism analysis
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Studying the genes expressed in samples of blood from young patients with cancer treated with ifosfamide may help doctors identify risk factors for kidney damage.

PURPOSE: This clinical trial is looking at the CYP3A5 gene to see if having the gene may be a risk factor for kidney damage in young patients with cancer treated with ifosfamide.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the CYP3A5 genotype in young patients with cancer who have received ifosfamide.
* To document renal function and nephrotoxicity on one occasion between 1 month and 5 years after completion of ifosfamide treatment.
* To determine the relationship between CYP3A5 genotype and ifosfamide nephrotoxicity.

Secondary

* To compare the measured glomerular filtration rate (GFR) (using a radioisotope clearance method) with that calculated using the Cole (weight and creatinine) model.

OUTLINE: This is a multicenter study.

Nephrotoxicity assessment is performed in patients who have not undergone prior assessment*.

NOTE: *Nephrotoxicity assessment is performed once between 1 month and 5 years after completion of ifosfamide chemotherapy.

All patients will undergo a single blood sample collection. DNA will be extracted from this sample and genotyped for the known functional polymorphisms in CYP3A5. The technique of restriction fragment length polymorphism (RFLP) will be used to detect any single nucleotide polymorphisms in CYP3A5.

DNA may be obtained from stored tumor samples from patients for whom the results of renal investigations are available, but for whom blood is not available for CYP3A5 genotyping.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Received ifosfamide before the age of 21 as part of treatment for cancer including, but not limited to, any of the following:

  * Ewing sarcoma
  * Rhabdomyosarcoma
  * Non-rhabdomyosarcoma soft tissue sarcoma
* No renal infiltration by tumor at any stage of illness
* May have been treated on one of the following clinical trials:

  * Euro-Ewing-Intergroup-EE99
  * SIOP-MMT-95

    * Patients who received CEV chemotherapy (carboplatin, epirubicin, and vincristine) on strategy 952 or 953 are not eligible
  * CCLG-EPSSG-NRSTS-2005
  * CCLG-EPSSG-RMS-2005

PATIENT CHARACTERISTICS:

* Clinically stable to undergo renal investigations
* No pre-existing renal impairment (glomerular or tubular) prior to treatment with ifosfamide
* No known nephrotoxicity for which nephrotoxic supportive treatment (aminoglycosides, amphotericin, acyclovir, cyclosporine, or tacrolimus) was a major contributory cause of renal damage

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from the acute non-renal toxicity of the last course of chemotherapy
* No other prior nephrotoxic chemotherapy (e.g., cisplatin, carboplatin, melphalan, or high-dose methotrexate)
* No prior radiotherapy to a field including the kidneys
* No prior removal of renal tissue
* No concurrent ifosfamide

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
CYP3A5 genotype
Renal function and nephrotoxicity
Relationship between CYP3A5 genotype and ifosfamide nephrotoxicity

SECONDARY OUTCOMES:
Comparison of measured glomerular filtration rate (GFR) with the Cole model

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Veal, Principal Investigator — University of Newcastle Upon-Tyne
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - University College Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales